CLINICAL TRIAL: NCT01919008
Title: Phase I Study of FK949E - Comparison of Pharmacokinetics Between FK949E 50 mg Tablets and FK949E 150 mg Tablets in Patients With Major Depressive Disorder
Brief Title: Comparison of Plasma Concentration Changes Between Two Types of Tablets of FK949E Administration to Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 6949-CL-0006
Record Dates: First submitted 2013-08-06; First posted 2013-08-08 (Estimated); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Major Depressive Disorder
Keywords: FK949E; Pharmacokinetics; Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (FK949E low dose tablet-first group) (Experimental): Days 1 and 2: One FK949E low dose tablet
  Days 3 to 6: Three FK949E low dose tablets
  Days 7 to 10: One FK949E high dose tablet
  Interventions: Drug: FK949E
- Group 2 (FK949E high dose tablet-first group) (Experimental): Days 1 and 2: One FK949E low dose tablet
  Days 3 to 6: One FK949E high dose tablet
  Days 7 to 10: Three FK949E low dose tablets
  Interventions: Drug: FK949E

INTERVENTIONS:
Drug: FK949E — Oral
  Other Names: extended release formulation of quetiapine

SUMMARY:
This study is to compare the pharmacokinetics of FK949E low dose tablets and FK949E high dose tablets in non-elderly patients with major depressive disorder. The safety of FK949E in the population was also evaluated.

DETAILED DESCRIPTION:
The objective of the study is to compare the pharmacokinetics of FK949E low dose tablets and FK949E high dose tablets in non-elderly patients with major depressive disorder in a 2 × 2 crossover design. The safety of FK949E in the population is also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients considered to be able to understand and follow subject requirements, as judged by the investigator/sub-investigator.
* Patients diagnosed with major depressive disorder according to the DSM-IV-TR by means of M.I.N.I.
* BMI: 17.6 (inclusive) to 26.4 (exclusive).

Exclusion Criteria:

* Current or past history of DSM-IV-TR Axis I disorder, except major depressive disorder, within the past 6 months before informed consent.
* Concurrent DSM-IV-TR Axis II disorder that is considered to greatly affect patient's current mental status.
* Current or past history of dependence of substances (other than caffeine and nicotine) or history of abuse or dependence of alcohol.
* Unable to suspend treatment with inducers or inhibitors of the drug-metabolizing enzyme, cytochrome P450 3A4 (CYP3A4), for 14 days before the screening assessment and throughout the study.
* Patients who could not use an appropriate contraception (condoms) during the study. Patients who were pregnant or lactating.
* Patients (carriers) with documented or suspected renal failure, hepatic failure, serious cardiac disease,

hepatitis B, hepatitis C, or acquired immunodeficiency syndrome (AIDS).

* Patients receiving treatment for hypertension, or patients with concurrent hypertension or unstable angina that may worsen with the study or may affect the study results based on the clinical judgment of the investigator/sub-investigator.
* Patients with concurrent hypotension (criterion for hypotension: a systolic blood pressure of less than 100 mmHg), or orthostatic hypotension
* Patients with a mean QTcF interval of ≥450 ms on a 12-lead ECG at the screening assessment
* Patients with the risk of torsades de pointe (e.g., those with a history of QT prolongation, those with familial long QT syndrome).
* Concurrent malabsorption syndrome, hepatic disease, or other conditions that may affect the absorption and/or metabolism of the study drug.
* Concurrent malignancy or history of cured malignancy within 5 years
* Current or past history of cerebrovascular disease or transient ischemic attack (TIA).
* Received electroconvulsive therapy within 90 days before the screening assessment

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2012-03-26 (Actual); Primary Completion 2012-06-22 (Actual); Study Completion 2012-06-22 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of unchanged quetiapine | For 24 hours after dosing
  Frequent blood sampling on Day 6 and Day 10
AUC24h (area under the curve for 24hr) of unchanged quetiapine | For 24 hours after dosing
  Frequent blood sampling on Day 6 and Day 10

SECONDARY OUTCOMES:
Trough value of plasma concentration of unchanged quetiapine | For 24 hours after dosing
  Frequent blood sampling on Day 6 and Day 10
t1/2 of plasma concentration of unchanged quetiapine | For 24 hours after dosing
  Frequent blood sampling on Day 6 and Day 10
Maximum plasma concentration (Cmax) of quetiapine metabolites | For 24 hours after dosing
  Frequent blood sampling on Day 6 and Day 10
AUC (area under the curve) of quetiapine metabolites | For 24 hours after dosing
  Frequent blood sampling on Day 6 and Day 10
trough value of plasma concentration of quetiapine metabolites | For 24 hours after dosing
  Frequent blood sampling on Day 6 and Day 10
tmax of plasma concentration of quetiapine metabolites | For 24 hours after dosing
  Frequent blood sampling on Day 6 and Day 10
t1/2 of plasma concentration of quetiapine metabolites | For 24 hours after dosing
  Frequent blood sampling on Day 6 and Day 10
Safety assessed by the incidence of adverse events, clinical tab tests, vital signs, 12-lead ECGs and physical exam | Up to Day 11

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (1):
- Kanto, Japan

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Fukushi R, Nomura Y, Katashima M, Komatsu K, Sato Y, Takada A. Approach to Evaluating QT Prolongation of Quetiapine Fumarate in Late Stage of Clinical Development Using Concentration-QTc Modeling and Simulation in Japanese Patients With Bipolar Disorder. Clin Ther. 2020 Aug;42(8):1483-1493.e1. doi: 10.1016/j.clinthera.2020.06.002. Epub 2020 Aug 11. PMID 32792252
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/hcp/study.aspx?ID=175